CLINICAL TRIAL: NCT03454334
Title: To Compare the Clinical Results of Different Multifocal Intraocular Lenses (IOLs) in Patients With Presbyopia or Cataracts
Brief Title: Visual Performance of Four Types of Multifocal Intraocular Lenses
Acronym: presbyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, farinaz doroodgar, Ophthalmologist, Shahid Beheshti University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShahedBU
Record Dates: First submitted 2018-01-25; First posted 2018-03-05 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2020-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Multifocal Intraocular Lenses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- AMO Tecnis Symfony (Active Comparator): Multifocal with extended range of vision, Diffractive, No Preloaded, Aspheric, +3.25 D near add and +2.17 D intermediate 6.0mm Hydrophilic
  -0.20
  Has nine diffractive steps, The proprietary achromatic technology corrects chromatic aberration. This creates improved contrast sensitivity.
  Interventions: Device: multifocal intraocular lens IOLs
- AcrySof ReSTOR (Alcon Laboratories) (Active Comparator): Multifocal ,Diffractive, +3.00D and for Near, Aspheric, Has 9 steps (rings), Light: 41% for far; 41% for near: 18% reflected (lost).
  6.0mm Silicone
  -0.10 Bifocal ,One piece,Blue filter ,Central diffractive region of 3.6_mm for near and distance vision ,Apodised ,peripheral refractive region is dedicated to distance vision
  Interventions: Device: multifocal intraocular lens IOLs
- AT Lisa tri (CarlZeiss Meditec AG) (Active Comparator): Trifocal, diffractive, +3.33 D near add and +1.66 D intermediate add at the IOL plane, aspheric (aberration correcting) Optic Diameter 6.0 mm Total Diameter 11.0 mm Haptic Angulation 0° Lens Design Single-piece, MICS Incision Size 1.8 mm Company Labeled A-Constant1 118.6 Diopter Range 0.0 to +32.0 D, 0.5 D increments ACD 5.32
  Interventions: Device: multifocal intraocular lens IOLs
- PanOptix(Alcon Laboratories) (Active Comparator): Trifocal,Difractive,+3.25D Near,+2.17 D intermediate 6.0mm hydrophobic
  -0.27 One piece ,aspheric , Focal 4.5 mm (15 diffractive zones)
  Interventions: Device: multifocal intraocular lens IOLs

INTERVENTIONS:
Device: multifocal intraocular lens IOLs — clinical outcome of different multifocal intraocular lenses (IOLs) in patients with presbyopia or cataracts

SUMMARY:
This investigation assessed the visual performance of presbyopia and cataract patients after bilateral implantation of 4 distinct sorts of multifocal IOLs: At lisa tri, PanOptix, ReSTOR, and Symfony. The clinical results demonstrated here were excellent for four groups, however, there were also differences in group ReSTOR, UCVA and BCVA for the intermediate and near of the other groups showed less vision also symphony group for far distance demonstrated less vision than other groups, which may be related to their design.Multifocal IOLs demonstrated very good technology and unquestionably have a place in refractive surgery, whether for clear lens extraction or cataracts.Patients can expect excellent outcomes and surgeons can expect patients to be very satisfied with surgical outcomes. Four groups multifocal lenses provided excellent distance, intermediate and near vision, but several measures indicated that the PanOptix and at lisa tri lens provided better vision in all distances. Spectacle independence was significantly higher with four groups. Multifocal IOL design might play a role in the postsurgical outcome, because better results were obtained with diffractive lenses. Although there were differences in the results of these four lenses in the study, all of the results were acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative BCVA (distance) more impacted than 20/40
* Glare VA test comes about worse than 20/40, or practically impairing dissensions about their vision.
* By reviewing and judging the researchers, individuals also had a potential need for visual acuity of 20/30 or better after surgery.
* Express a want for multifocal vision, and be ready and ready to conform to the investigation necessities

Exclusion Criteria:

* Excluded from entry were subjects with regular astigmatism greater than 1.5 D or irregular astigmatism.
* Large pupil
* Corneal transplant surgery or previous glaucoma-filtering,
* A history of retinal detachments.
* Also excluded were patients with other clinically non-cataract ocular abnormality (e.g. chronic drug-induced miosis,
* Endothelial disease
* Iris neovascularization, and amblyopia)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-08-11 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity | 4 years
  mean postoperative contrast sensitivity in logarithmic scale under binocular mesopic and photopic conditions. There was no significant difference in the values obtained between at lisa tri and PanOptix at spatial frequencies of 1 cpd and 3, 6, 12, 18 cpd. Eyes with the PanOptix and at lisa tri IOL showed better contrast sensitivity than ReSTOR and Symfony at spatial frequencies of 1, 3, 6 cpd (P<0.001) in photopic and mesopic conditions. The curves achieved with monocular vision were equivalent with binocular vision that was achieved.